CLINICAL TRIAL: NCT02270203
Title: LOIS: Long-Term Follow-Up in INSITE/SIFI
Acronym: LOIS
Status: Completed | Type: Observational
Sponsor: SI-BONE, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 300244
Record Dates: First submitted 2014-10-16; First posted 2014-10-21 (Estimated); Last update posted 2019-08-06 (Actual); Status verified 2019-08

CONDITIONS: Degenerative Sacroilitis; Sacroiliac Joint Disruption
Keywords: si joint; si joint injury; si joint treatment; si joint inflammation; si joint problems; si joint symptoms; hypermobile joint; si joint arthritis; si joint pain treatment; inflamed si joint; si joint sclerosis; locked si joint; si joint injuries; si joint disease; si joint infection; sacroiliac joint pelvic pain; sacroiliac joint arthritis treatment; si joint pain; si joint injections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Radiation: Pelvic CT at 5 years post-op — Pelvic CT at 5 years post-op

SUMMARY:
The purpose of this study is to evaluate the long term safety and effectiveness of SI joint fusion using the iFuse Implant System in patients with degenerative sacroiliitis (DS) and/or sacroiliac joint disruptions (SD).

Study Design: This study is extended follow-up from two ongoing multicenter prospective US clinical trials. All participants have already undergone the surgical procedure of interest (SI joint fusion with iFuse Implant System). The two ongoing trials are:

* SIFI:( Sacroiliac Joint Fusion with iFuse Implant System) a single-arm trial of patients with degenerative sacroiliitis or sacroiliac joint disruption who underwent iFuse placement, and
* INSITE(Investigation of Sacroiliac Fusion Treatment): a randomized clinical trial of the same patient population who underwent either non-surgical treatment or iFuse placement

ELIGIBILITY:
Inclusion Criteria:

1. Patient enrolled and treated in SIFI or patient initially randomized to iFuse and treated in INSITE. Note: Patient may be in the initial follow up period associated with SIFI or INSITE at the same time they consent for this study and "extend" their post-operative follow up.
2. Patient has signed study-specific LOIS informed consent form.
3. Patient has the necessary mental capacity to participate and is physically able to comply with study protocol requirements.

Exclusion Criteria:

1. Treated with iFuse as a "crossover" in INSITE.
2. Currently pregnant or planning pregnancy within 5 years of iFuse Implant.
3. Patient is a prisoner or a ward of the state.
4. Known or suspected active drug or alcohol abuse.
5. Inadequately treated psychiatric illness (e.g., schizophrenia, major depression, personality disorders) that could interfere with study participation.
6. Unwilling to perform the long-term follow up requirements of this study.
7. Patient has any condition that could substantially prevent long-term follow-up.
8. Unwilling to return to site at pre-specified study visits.

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects with degenerative sacroiliitis or sacroiliac joint disruption who underwent iFuse placement.
Sampling Method: Non-Probability Sample
Enrollment: 103 (Actual)
Dates: Start 2014-10; Primary Completion 2019-07 (Actual); Study Completion 2019-07 (Actual)

PRIMARY OUTCOMES:
Subject Success | 3 years on LOIS (5 years post-op)
  Composite endpoint of success defined as improvement in VAS (Visual Analog Scale) recorded at SIFI or INSITE Baseline VAS back pain score by ≥20 mm; Absence of device-related SAE (Serious Adverse Events) ; Absence of neurological worsening related to the sacral spine,& Absence of surgical re-intervention on the target SI joint(s).
Radiographic (CT) apposition of bone to sacral and iliac sides of implant | 3 years on LOIS (5 years post-op)
  Proportion of subjects (with CT) who had at least 30% apposition of bone to sacral and iliac sides in at least 2 of 3 iFuse implants.

SECONDARY OUTCOMES:
VAS (Visual Analog Scale) | 3 years on LOIS (5 years post-op)
  Improvement in VAS (Visual Analog Scale), SI joint pain at follow-up visits.
Oswestry Disability Index (ODI) Questionnaire | 3 years on LOIS (5 years post-op)
  Improvement in Oswestry Disability Index (ODI) at follow-up visits.
Improvement in quality of life (QOL) | 3 years on LOIS (5 years post-op)
  Improvement in quality of life as measure by EQ-5D Questionnaire at follow-up visits.
non-working subjects returning to work | 3 years on LOIS (5 years post-op)
  Proportion of non-working subjects who return to work
CT scans showing bridging bone | 3 years on LOIS (5 years post-op)
  Proportion of CT scans that show bridging bone across the SI joint at 5 years post-operatively
SAE (Serious Adverse Events) occurrence rate | 3 years on LOIS
  Occurrence rate of serious adverse events.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Cher, MD, Study Director — SI-BONE, Inc.
Locations (12):
- United States (12):
  - Yale University School of Medicine, New Haven, Connecticut
  - Regenerative Orthopaedics and Spine Institute, Stockbridge, Georgia
  - Orthopaedic Center of Southern Illinois, Mount Vernon, Illinois
  - Bluegrass Orthopaedics & Hand Care, Lexington, Kentucky
  - Columbia Orthopaedic Group, Columbia, Missouri
  - Oklahoma Center for Spine & Pain Solutions, Oklahoma City, Oklahoma
  - Allegheny Medical Center, Pittsburgh, Pennsylvania
  - MUSC, Charleston, South Carolina
  - Precision Spine Care, Tyler, Texas
  - Overlake Hospital Medical Center, Bellevue, Washington
  - Aurora Research Institute, Green Bay, Wisconsin
  - Integrated Spine Care, Wauwatosa, Wisconsin

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Darr E, Cher D. Four-year outcomes after minimally invasive transiliac sacroiliac joint fusion with triangular titanium implants. Med Devices (Auckl). 2018 Aug 29;11:287-289. doi: 10.2147/MDER.S179003. eCollection 2018. PMID 30214322